CLINICAL TRIAL: NCT04385966
Title: Diaphragmatic Paralysis After Interscalene Brachial Plexus Block: A Randomized, Double-blinded, Unicenter and Controlled Clinical Trial to Reduce the Dose of Levobupivacaine 0,25% 20 ml to 10 ml Undergoing Arthroscopic Shoulder Surgery
Brief Title: Diaphragmatic Paralysis Comparison Between Local Anesthetic Volumen Doses After Interscalene Block
Acronym: REDOLEV-2019
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: REDOLEV-2019
Record Dates: First submitted 2020-04-16; First posted 2020-05-13 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2021-08

CONDITIONS: Diaphragmatic Paralysis; Brachial Plexus Block
Keywords: Diaphragmatic Paralysis; Interscalene Brachial Plexus Block; Ultrasound; Postoperative pain; Arthroscopic shoulder surgery.
MeSH Terms: conditions — Respiratory Paralysis; Pain, Postoperative | interventions — Levobupivacaine

STUDY DESIGN:
Intervention Model Description: The REDOLEV study is a randomized, comparative, prospective, unicenter, double-blind, two-arm and controlled Clinical trial (RCT).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After randomization, only Interscalene Block performer staff will know which intervention group is assigned to the participants. Spirometry and ultrasound assessments will be conducted by only one blinded anesthesiologist of Assessment staff who will not be communicated to IBPB staff. Recruitment and Assessment staff and participants will not be allowed to receive any information about the group allocation. Study unblinding will occur when every ultrasound and Spirometry assessments have been completed after 24-hour follow-up postoperative closeout. After follow-up finished, every study data will figure in the patient medical record. Code breaks should occur only in exceptional circumstances when knowledge of the actual treatment is absolutely essential for further management of the patient as an allergy episode. The Research staff will be encouraged to maintain the blind as far as possible. Unblinded IBPB staff will manage the emergency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Volume Dose (Active Comparator): 24 patients will be included in the Standard Volume Dose arm. 20 ml Levobupivacaine Hydrochloride 2.5 MG/ML will be administered in the Interscalene brachial plexus block before the arthroscopic shoulder surgery.
  Interventions: Procedure: Interscalene brachial plexus block; Drug: Levobupivacaine Hydrochloride 2.5 MG/ML
- Low Volume Dose (Experimental): 24 patients will be included in the Low Volume Dose arm. 10 ml Levobupivacaine Hydrochloride 2.5 MG/ML will be administered in the Interscalene brachial plexus block before the arthroscopic shoulder surgery.
  Interventions: Procedure: Interscalene brachial plexus block; Drug: Levobupivacaine Hydrochloride 2.5 MG/ML

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — Interscalene brachial plexus block is a locorregional anaesthesia technique which is indicated in shoulder and upper arm surgery. The goal of this block is to place the needle in the tissue space between the anterior and middle scalene muscles and inject local anesthetic until the spread around the brachial plexus is documented by ultrasound.
  Other Names: MeSH Unique ID: D065527; CIE-10 code 3E0T3CZ; Interscalene block
Drug: Levobupivacaine Hydrochloride 2.5 MG/ML — Levobupivacaine Hydrochloride 2.5 MG/ML is an anesthestic product intended for epidural, intradural and perineural administration. Levobupivacaine is chemically described as (S)-l-butyl-2-piperidylformo-2',6'-xylidide hydrochloride. It is a white crystalline powder with a molecular formula of C18H28N2O. HCl, with a molecular weight 324.9.
  FDA approval: NDA-20997 (1999).
  Other Names: Chirocaine® 2.5 MG/ML

SUMMARY:
Arthroscopic shoulder surgery involves dynamic and severe postoperative pain. Interscalene brachial plexus block (IBPB) provides adequate analgesia but the spread of local anaesthetics administered causes a phrenic nerve block which entrains a non-negligible incidence of Hemidiaphragmatic paralysis acute (HDPA).

This is a comparative, prospective, Unicenter, double-blind, two-arm, randomized and controlled clinical trial. 48 patients will be included.

This RCT would demonstrate a low volume dose IBPB decrease the HDPA after IBPB in patients undergoing SAS, by using spirometry and ultrasound and it will not provide inferior postoperative analgesia according to opioid requirements of postoperative PCA in comparison to standard volume dose used in current practice.

DETAILED DESCRIPTION:
Arthroscopic shoulder surgery involves dynamic and severe postoperative pain. Interscalene brachial plexus block (IBPB) provides adequate analgesia but the spread of local anaesthetics administered causes a phrenic nerve block which entrains a non-negligible incidence of Hemidiaphragmatic paralysis acute (HDPA).

The primary study objective is to determine the HDPA diagnosed by using diaphragmatic thickness index in Ultrasound (US) after Low Volume (10 mL) versus Standard Volume (20 mL) of Levobupivacaine 0,25% for IBPB. Secondary end-points are 1) HDPA diagnosed by using FVC and FEV1 in spirometry, 2) HDPA diagnosed by using diaphragmatic excursion in US, 3) postoperative pain regarding time to first analgesic consumption and 24-hour cumulative total consumption of Patient-controlled analgesia (PCA) pump of Morphine IV and (4) postoperative harms between two trial-arms.

This study is a comparative, prospective, Unicenter, double-blind and two-arm RCT. 48 patients will be included.

This RCT would demonstrate a low volume dose IBPB decrease the HDPA after IBPB in patients undergoing SAS, by using spirometry and ultrasound and it will not provide inferior postoperative analgesia according to opioid requirements of postoperative PCA in comparison to standard volume dose used in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years.
* ASA I-III.
* Scheduled for shoulder arthroscopic shoulder surgery and interscalene brachial plexus block.

Exclusion Criteria:

* Age <18 and >80 years.
* Pregnancy.
* Exclusión to perform IBPB or spirometry.
* Allergy to amide group local anaesthetics, opioids or nonsteroidal anti-inflammatory drugs.
* Background of Pulmonary diseases (chronic obstructive pulmonary disease (COPD) and moderate, severe or not well-controlled asthma), diaphragmatic paralysis or neurological disease with diaphragmatic dysfunction, brachial plexus neuropathy or chronic opioid consumption (more than 3-months consumption or more than oral Morphine 1 mg 1-month).
* Coagulation disorders (INR>3, TTPA > 35 y AP <50%).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Diaphragmatic Thickness Ratio at 4 hours | Before (Baseline) and 4-hour after interscalene brachial plexus block
  The primary outcome is the difference in the proportion of patients with Hemidiaphragmatic paralysis acute (HDPA) according to diaphragmatic thickness ratio (DTR) in ultrasounds between the Treatment and Control groups. DTR will be the result of Inspiratory Diaphragmatic Thickness and Expiratory Diaphragmatic Thickness. The ratio will be defined by DTR=IDT/EDT. HDPA after IBPB at 4 hours will be diagnosed with a DTR<1.2.

SECONDARY OUTCOMES:
Change from Baseline FVC at 4 hours and 24 hours | Before (Baseline), 4-hour and 24-hour after interscalene brachial plexus block
  This secondary outcome is the difference in the proportion of patients with Hemidiaphragmatic paralysis acute (HDPA) according to Forced Vital Capacity (FVC) in spirometry. HDPA will be diagnosed with a CVF diminution of >20%.
Change from Baseline FEV1 at 4 hours and 24 hours | Before (Baseline), 4-hour and 24-hour after interscalene brachial plexus block
  This secondary outcome is the difference in the proportion of patients with Hemidiaphragmatic paralysis acute (HDPA) according to forced expiratory volume in one second (FEV1) in spirometry. HDPA will be diagnosed with a FEV1 diminution of >20%.
Change from Baseline Diaphragmatic excursion at 4 hours and 24 hours | Before (Baseline), 4-hour and 24-hour after interscalene brachial plexus block
  This secondary outcome is the difference in the proportion of patients with Hemidiaphragmatic paralysis acute (HDPA) according to Diaphragmatic excursion expressed as number of intercostal spaces and motion type. HDPA will be diagnosed with a reduction of >25% number of intercostal spaces or a paradoxal or nule diaphragmatic motion.
Postoperative IV morphine consumption | From 4-hour to 24-hour after interscalene brachial plexus block
  This secondary outcome is the postoperative 24-hour cumulative IV morphine consumption (mg) of Patient controlled analgesia (PCA) pump.
Postoperative time to first analgesic consumption | From 4-hour to 24-hour after interscalene brachial plexus block
  This secondary outcome is the time to first analgesic consumption (minutes) of Patient controlled analgesia (PCA) pump.
Incidence and frequency of Serious Adverse Events (SAE) | From performing the interscalene brachial plexus block to finish the 24-hour postoperative follow-up
  This secondary outcome is the incidence, frequency and severity of Serious Adverse Events (SAE) as assessed by CTCAE v4.0 in the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Pablo O Forniés, MD, Principal Investigator — Hospital Miguel Servet
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be available on file in storage and on the Internet (URL undecided yet) after finishing the data collection for 25 years at the participating site.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting in February 2021 for 25 years.
Access Criteria: * To contact to Study Principal Investigator.
  * To provide to Study Principal Investigator a request to explain the reason to access to IPD study.

REFERENCES:
- [Background] Lopez Escarraga VM, Dubos Espana K, Castillo Bustos RH, Peidro L, Sastre S, Sala-Blanch X. Diaphragmatic thickness ratio (inspiratory/expiratory) as a diagnostic method of diaphragmatic palsy associated with interescalene block. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Feb;65(2):81-89. doi: 10.1016/j.redar.2017.09.008. Epub 2017 Nov 7. English, Spanish. PMID 29126611
- [Background] Urmey WF, McDonald M. Hemidiaphragmatic paresis during interscalene brachial plexus block: effects on pulmonary function and chest wall mechanics. Anesth Analg. 1992 Mar;74(3):352-7. doi: 10.1213/00000539-199203000-00006. PMID 1539813
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Thackeray EM, Swenson JD, Gertsch MC, Phillips KM, Steele JW, Burks RT, Tashjian RZ, Greis PE. Diaphragm function after interscalene brachial plexus block: a double-blind, randomized comparison of 0.25% and 0.125% bupivacaine. J Shoulder Elbow Surg. 2013 Mar;22(3):381-6. doi: 10.1016/j.jse.2012.06.011. Epub 2012 Sep 1. PMID 22947235
- [Background] Stundner O, Meissnitzer M, Brummett CM, Moser S, Forstner R, Kokofer A, Danninger T, Gerner P, Kirchmair L, Fritsch G. Comparison of tissue distribution, phrenic nerve involvement, and epidural spread in standard- vs low-volume ultrasound-guided interscalene plexus block using contrast magnetic resonance imaging: a randomized, controlled trial. Br J Anaesth. 2016 Mar;116(3):405-12. doi: 10.1093/bja/aev550. PMID 26865133
- [Derived] Oliver-Fornies P, Ortega Lahuerta JP, Gomez Gomez R, Gonzalo Pellicer I, Oliden Gutierrez L, Vinuales Cabeza J, Gallego Ligorit L, Orellana Melgar CE. Diaphragmatic paralysis, respiratory function, and postoperative pain after interscalene brachial plexus block with a reduced dose of 10 ml levobupivacaine 0.25% versus a 20 ml dose in patients undergoing arthroscopic shoulder surgery: study protocol for the randomized controlled double-blind REDOLEV study. Trials. 2021 Apr 19;22(1):287. doi: 10.1186/s13063-021-05216-6. PMID 33874993

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT04385966/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT04385966/ICF_001.pdf